CLINICAL TRIAL: NCT02917395
Title: Evaluate the Efficacy of Disopyramide Therapy in Hypertrophic Obstructive Cardiomyopathy Patients; Comparison of Two Echocardiography Based Methods: Global Longitudinal Strain vs. Left Ventricle Ejection Fraction
Brief Title: Evaluate the Efficacy of Disopyramide Therapy in Hypertrophic Obstructive Cardiomyopathy Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Idit Yedidya, Head of echo lab- hashron campus in Rabin medical center, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 0538-16-RMC
Record Dates: First submitted 2016-09-27; First posted 2016-09-28 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Cardiomyopathy
Keywords: hypertrophic cardiomyopathy, disopyramide,
MeSH Terms: conditions — Cardiomyopathies; Cardiomyopathy, Hypertrophic | interventions — Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- echo (Experimental): Population study- patients with obstructive hypertrophic cardiomyopathy that are treated with disopyramide.
  Tow echo examination, few hours apart, that includes strain rate will be done to each patient. The first, after taking the regular medical treatment excluding disopyramide and the last one after taking the disopyramide.
  Interventions: Device: echocardiography

INTERVENTIONS:
Device: echocardiography — Tow echo examination, few hours apart, that includes strain rate will be done to each patient. The first, after taking the regular medical treatment excluding disopyramide and the last one after taking the disopyramide.

SUMMARY:
Population study- patients with obstructive hypertrophic cardiomyopathy that are treated with disopyramide.

Tow echo examination, few hours apart, that includes strain rate will be done to each patient. The first, after taking the regular medical treatment excluding disopyramide and the last one after taking the disopyramide.

DETAILED DESCRIPTION:
Tow echo examination, few hours apart, that includes strain rate will be done to each patient. The first, after taking the regular medical treatment excluding disopyramide and the last one after taking the disopyramide.

ELIGIBILITY:
Inclusion Criteria:

* hypertrophic cardiomyopathy that treated with disopyramid

Exclusion Criteria:

* pregnancy
* pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-01 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Tow echo examination, few hours apart, that includes strain rate will be done to each patient. The first, after taking the regular medical treatment excluding disopyramide and the last one after taking the disopyramide | 2-3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Idit Yedidya, MD, Principal Investigator — Rabin Medical Center

IPD SHARING:
Plan to Share IPD: Undecided